CLINICAL TRIAL: NCT05827757
Title: Single-group, Open-label, Phase I / II Clinical Trial: Evaluating the Safety and Efficacy of Autologous Adipose Tissue-derived Mesenchymal Stem Cell Transplantation on Proinflammatory Cytokines and Cytokines Balance in Inflammaging (Ageing-related Low-grade Inflammation) Patients.
Brief Title: Evaluating the Safety and Efficacy of Autologous Adipose Tissue-derived Mesenchymal Stem Cell Transplantation on Proinflammatory Cytokines and Anti-inflammatory Cytokines on Ageing-related Low-grade Inflammation Patients.
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: DNA International Hospital (Other)
Collaborators: University of Science Ho Chi Minh City (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 1690/QĐ-BYT
Record Dates: First submitted 2020-10-13; First posted 2023-04-25 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-10

CONDITIONS: Aging Problems; Aging; Chronic Inflammation
Keywords: Ageing-related low-grade inflammation;; inflammaging;; aging

STUDY DESIGN:
Intervention Model Description: Evaluating the Safety and Efficacy of Autologous Adipose Tissue-derived Mesenchymal Stem Cell Transplantation on Proinflammatory Cytokines and Anti-inflammatory Cytokines on Ageing-related Low-grade Inflammation Patients.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MSC transplantation (Experimental): Transplant 100 million MSCs
  Interventions: Biological: autologous adipose-derived mesenchymal stem cell transplantation

INTERVENTIONS:
Biological: autologous adipose-derived mesenchymal stem cell transplantation — Transplant 100 million autologous adipose-derived mesenchymal stem cells at Day 0 and Day 90

SUMMARY:
Single-group, open-label, phase I / II clinical trial: Evaluation of the safety of autologous adipose tissue-derived mesenchymal stem cell transplantation in inflammaging (Ageing-related low-grade inflammation) patients.

DETAILED DESCRIPTION:
The proposed study is a single-group, open-label, phase I / II clinical trial in which the patients will be treated with two doses (100 million i.v) of autologous adipose tissue-derived mesenchymal stem cell transplantation.

This study aims to evaluate the safety and efficiency of autologous adipose tissue-derived mesenchymal stem cell transplantation in inflammaging (Ageing-related low-grade inflammation) patients. The inflammaging-patients are who have cytokine increasing (IL6 and TNF alfa)

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patient, age 40 to 64 years.
2. The inflammatory aging patient as defined in the protocol as TNF alpha or IL6 at the time of screening was higher than the 95% healthy percentile value declared by the test system manufacturer.
3. Have at least 2 of the 3 following diseases:

   * Diabetes type II
   * Dyslipidemia
   * Obesity [The diagnosis and determination of accompanying diseases (Diabetes, Dyslipidemia, Obesity) will be carried out according to the general guidance of the MOH Vietnam].
4. Patients are using stable drugs for co-infection (diabetes mellitus, dyslipidemia, obesity) stably in the past 3 months.
5. Agree to participate in research and agree to comply with the research examination and evaluation process.

Exclusion Criteria:

1. Patients with a blood-clotting disorder or hemophilia
2. Patients with severe heart failure
3. Acute respiratory pathology at the time of screening
4. Patients with cancer or other acute illness need treatment.
5. Patients with a history of allergy to anesthetics, anesthesia, and antibiotics
6. Patients are planning to participate in another clinical trial while participating in the study
7. There are other conditions or circumstances in which it is difficult for researchers to ensure adherence to treatment in the judgment of researchers.

Ages: 40 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2020-04-28 (Actual); Primary Completion 2025-04-13 (Estimated); Study Completion 2025-04-13 (Estimated)

PRIMARY OUTCOMES:
The safety and toleration of stem cell infusion | Study recruirement day 0
  Assess the safety and tolerance of autologous adipose-derived mesenchymal stem cell transplantation in patients with inflammatory aging. During the entire duration of the study, the likelihood of adverse event occurrence and adverse event effects related or unrelated to stem cell infusion will be reported according to Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
The safety and toleration of stem cell infusion | Day 90
  Assess the safety and tolerance of autologous adipose-derived mesenchymal stem cell transplantation in patients with inflammatory aging. During the entire duration of the study, the likelihood of adverse event occurrence and adverse event effects related or unrelated to stem cell infusion will be reported according to Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
The safety and toleration of stem cell infusion | Study endpoint at day 180
  Assess the safety and tolerance of autologous adipose-derived mesenchymal stem cell transplantation in patients with inflammatory aging. During the entire duration of the study, the likelihood of adverse event occurrence and adverse event effects related or unrelated to stem cell infusion will be reported according to Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.

SECONDARY OUTCOMES:
The change of proinflammatory cytokines after stem cell transplantation in patients | Day 0, Day 90 and Day 180
  The measurement of proinflammatory cytokines concentration in patients peripheral blood such as IL-1α (pg/ml), IL-1β (pg/ml), TNF-α (pg/ml), TNF-β (pg/ml), IL-6 (pg/ml), IL-11 (pg/ml), IL-18 (pg/ml), IFN-γ (pg/ml) at day 0, 90, and 180 after stem cell infusion.
  During the study period, the variation of cytokine levels in individual patients revealed the results.
The change of anti-inflammatory cytokines after stem cell transplantation in patients | Day 0, Day 90 and Day 180
  At day 0, 90, and 180 after stem cell infusion, the concentration of anti-inflammatory cytokines such as IL - 4 (pg/ml), IL-10 (pg/ml), EGF (pg/ml), and MCP-1 (pg/ml) in the peripheral blood of patients is measured.
  During the study period, the variation of cytokine levels in individual patients revealed the results.
The influence of stem cell transplantation on thechange of the ratio of pro-inflammatory to anti-inflammatory cytokines | Day 0, Day 90 and Day 180
  The ratio of pro-inflammatory cytokines to anti-inflammatory cytokines will be used to assess the inflammation balance. The ratios from baseline were compared to three and six months after stem cell infusion such as IL-4/IL-10, IL-1/IL-10, IL-6/IL-10, and IL-1/EGF will be reported.

CONTACTS AND LOCATIONS:
Locations (1):
- DNA International Hospital, Ho Chi Minh City, District 05, Vietnam

REFERENCES:
- [Derived] Nguyen NT, Phan HT, Le PM, Nguyen LT, Do TT, Phan TT, Van Le T, Dang TM, Phan CL, Dang TT, Truong NH. Safety and efficacy of autologous adipose tissue-derived stem cell transplantation in aging-related low-grade inflammation patients: a single-group, open-label, phase I clinical trial. Trials. 2024 May 8;25(1):309. doi: 10.1186/s13063-024-08128-3. PMID 38715140